CLINICAL TRIAL: NCT02961647
Title: Invasive Hemodynamic Stress Test in Symptomatic and Asymptomatic Mitral Regurgitation
Brief Title: Hemodynamic Stress Test in Severe Mitral Regurgitation (HEMI)
Acronym: HEMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Heart Foundation (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Rine Bakkestrøm, Principal investigator, Odense University Hospital
Other Study IDs: A5130
Record Dates: First submitted 2016-10-06; First posted 2016-11-11 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Mitral Valve Regurgitation
Keywords: Hemodynamic stress test; Surgical intervention
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood and tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Asymptomatic patients: Patients with asymptomatic severe mitral valve regurgitation not undergoing surgical repair of the valve.
- Symptomatic patients: Patients with symptomatic severe mitral valve regurgitation undergoing surgical repair of the valve.
  Interventions: Procedure: Mitral valve repair

INTERVENTIONS:
Procedure: Mitral valve repair — The intervention is NOT related to the study design. It is a description of patients undergoing surgery vs. not undergoing surgery and this decision is made according to current guidelines (patients are not randomized).
  Groups: Symptomatic patients

SUMMARY:
The preferred treatment of organic mitral regurgitation (MR) is mitral valve repair. Optimally this should be timed so late that it commensurate with the risk of surgery and before irreversibly damage of the heart and pulmonary vessels. The aim is to obtain an understanding of the differences between the symptomatic and asymptomatic patient.

The study will test

A: Symptomatic organic MR is characterized by higher filling pressure, and higher stroke work during physical strain compared with asymptomatic MR.

B: The extent of myocardial fibrosis is associated with filling pressure and cardiac index 1 year after mitral valve repair.

C: Filling pressure can be estimated non-invasively by echocardiography. To test this 40 patients with asymptomatic MR and 40 symptomatic will undergo a stress echocardiography with simultaneous echocardiography and invasive measurement of central hemodynamics. In addition a pulmonary function test and cardiac MRI will be performed.

DETAILED DESCRIPTION:
Background

Degenerative mitral valve disease is the most common cause of organic mitral regurgitation in the Western World. The preferred treatment of organic mitral regurgitation is mitral valve repair. Optimally this should be timed so late that it commensurate with the risk of surgery and before irreversibly damage of the heart and pulmonary vessels. According to the current guidelines mitral valve surgery is indicated in symptomatic patients with severe MR or in presence of known risk factors. The optimal timing of surgery is still controversial in the asymptomatic patients without risk factors.

The overall aim of the present study is to obtain a better understanding of the central hemodynamics at rest and during physical exercise in both symptomatic and asymptomatic patients with organic mitral regurgitation, the relation to neurohormonal activation and myocardial fibrosis, and to identify noninvasive echocardiographic measures suitable for estimation of this.

A epidemiologic sub-study aims to asses whether MR is associated with inherence, as familial clustering of mitral regurgitation earlier has been suggested based only mainly on small observational studies, and case reports.

Methods

The study will test

A: Symptomatic organic MR is characterized by higher filling pressure, and higher stroke work during physical strain compared with asymptomatic MR.

B: The extent of myocardial fibrosis is associated with filling pressure and cardiac index 1 year after mitral valve repair.

C: Filling pressure can be estimated non-invasively by echocardiography.

To test this 40 patients with asymptomatic MR and 40 patients with symptomatic MR will undergo a stress echocardiography with simultaneous echocardiography and invasive measurement of central hemodynamics. In symptomatic patients that undergo surgery, the examination will be repeated 1 year after the surgical mitral valve repair.

In addition pulmonary function test, maximal oxygen consumption test and cardiac MRI will be performed.

The Danish Twin Registry and The Danish National Patient Registry will be used to identify twins with MR. The hypothesis is that the concordance rate is higher in monozygotic twins compared to dizygotic twins.

ELIGIBILITY:
Inclusion Criteria:

* Organic mitral valve regurgitation with effective regurgitation orifice (ERO)>0.3 cm2
* Age > 18 years
* Left ventricular ejection fraction (LVEF) > 60% assessed by echocardiography
* Signed informed consent

Exclusion Criteria:

* Poor echocardiographic window
* Inability to perform bicycle exercise testing
* Ischemic or functional (secondary) mitral valve regurgitation
* Chronic atrial fibrillation/flutter
* Hemodynamic significant aortic valve disease assessed by echocardiography.
* Treatment with oral anticoagulants

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the research project the investigators will examine 80 patients with severe MR, of which 40 do not experience symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Pulmonary artery wedge pressure | One year after mitral valve replacement

SECONDARY OUTCOMES:
Extent of myocardial fibrosis | One year after mitral valve replacement
Maximal oxygen consumption | One year after mitral valve replacement

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Møller, Professor, Principal Investigator — Department of Cardiology, Odense University Hospital
Locations (1):
- Department of Cardiology, Odense University Hospital, Odense, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS); Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Iung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M. Guidelines on the management of valvular heart disease (version 2012). Eur Heart J. 2012 Oct;33(19):2451-96. doi: 10.1093/eurheartj/ehs109. Epub 2012 Aug 24. No abstract available. PMID 22922415
- [Background] Bonow RO. Chronic mitral regurgitation and aortic regurgitation: have indications for surgery changed? J Am Coll Cardiol. 2013 Feb 19;61(7):693-701. doi: 10.1016/j.jacc.2012.08.1025. Epub 2012 Dec 19. PMID 23265342
- [Background] Enriquez-Sarano M, Avierinos JF, Messika-Zeitoun D, Detaint D, Capps M, Nkomo V, Scott C, Schaff HV, Tajik AJ. Quantitative determinants of the outcome of asymptomatic mitral regurgitation. N Engl J Med. 2005 Mar 3;352(9):875-83. doi: 10.1056/NEJMoa041451. PMID 15745978
- [Background] Suri RM, Vanoverschelde JL, Grigioni F, Schaff HV, Tribouilloy C, Avierinos JF, Barbieri A, Pasquet A, Huebner M, Rusinaru D, Russo A, Michelena HI, Enriquez-Sarano M. Association between early surgical intervention vs watchful waiting and outcomes for mitral regurgitation due to flail mitral valve leaflets. JAMA. 2013 Aug 14;310(6):609-16. doi: 10.1001/jama.2013.8643. PMID 23942679
- [Background] Naji P, Griffin BP, Asfahan F, Barr T, Rodriguez LL, Grimm R, Agarwal S, Stewart WJ, Mihaljevic T, Gillinov AM, Desai MY. Predictors of long-term outcomes in patients with significant myxomatous mitral regurgitation undergoing exercise echocardiography. Circulation. 2014 Mar 25;129(12):1310-9. doi: 10.1161/CIRCULATIONAHA.113.005287. Epub 2014 Jan 6. PMID 24396041
- [Background] Magne J, Mahjoub H, Pibarot P, Pirlet C, Pierard LA, Lancellotti P. Prognostic importance of exercise brain natriuretic peptide in asymptomatic degenerative mitral regurgitation. Eur J Heart Fail. 2012 Nov;14(11):1293-302. doi: 10.1093/eurjhf/hfs114. Epub 2012 Jul 10. PMID 22782970
- [Background] Ersboll M, Valeur N, Mogensen UM, Andersen MJ, Moller JE, Velazquez EJ, Hassager C, Sogaard P, Kober L. Prediction of all-cause mortality and heart failure admissions from global left ventricular longitudinal strain in patients with acute myocardial infarction and preserved left ventricular ejection fraction. J Am Coll Cardiol. 2013 Jun 11;61(23):2365-73. doi: 10.1016/j.jacc.2013.02.061. Epub 2013 Apr 3. PMID 23563128
- [Background] Witkowski TG, Thomas JD, Debonnaire PJ, Delgado V, Hoke U, Ewe SH, Versteegh MI, Holman ER, Schalij MJ, Bax JJ, Klautz RJ, Marsan NA. Global longitudinal strain predicts left ventricular dysfunction after mitral valve repair. Eur Heart J Cardiovasc Imaging. 2013 Jan;14(1):69-76. doi: 10.1093/ehjci/jes155. Epub 2012 Jul 29. PMID 22848021
- [Background] Dalsgaard M, Kjaergaard J, Pecini R, Iversen KK, Kober L, Moller JE, Grande P, Clemmensen P, Hassager C. Left ventricular filling pressure estimation at rest and during exercise in patients with severe aortic valve stenosis: comparison of echocardiographic and invasive measurements. J Am Soc Echocardiogr. 2009 Apr;22(4):343-9. doi: 10.1016/j.echo.2009.01.007. Epub 2009 Mar 9. PMID 19269785
- [Background] Andersen MJ, Ersboll M, Axelsson A, Gustafsson F, Hassager C, Kober L, Borlaug BA, Boesgaard S, Skovgaard LT, Moller JE. Sildenafil and diastolic dysfunction after acute myocardial infarction in patients with preserved ejection fraction: the Sildenafil and Diastolic Dysfunction After Acute Myocardial Infarction (SIDAMI) trial. Circulation. 2013 Mar 19;127(11):1200-8. doi: 10.1161/CIRCULATIONAHA.112.000056. Epub 2013 Feb 13. PMID 23406672
- [Derived] Andersen MJ, Wolsk E, Bakkestrom R, Christensen N, Carter-Storch R, Omar M, Dahl JS, Frederiksen PH, Borlaug B, Gustafsson F, Hassager C, Moller JE. Pressure-flow responses to exercise in aortic stenosis, mitral regurgitation and diastolic dysfunction. Heart. 2022 Nov 10;108(23):1895-1903. doi: 10.1136/heartjnl-2022-321204. PMID 36356959
- [Derived] Bakkestrom R, Banke A, Pecini R, Irmukhamedov A, Nielsen SK, Andersen MJ, Borlaug BA, Moller JE. Cardiac remodelling and haemodynamic characteristics in primary mitral valve regurgitation. Open Heart. 2018 Dec 16;5(2):e000919. doi: 10.1136/openhrt-2018-000919. eCollection 2018. PMID 30613416
- [Derived] Bakkestrom R, Banke A, Christensen NL, Pecini R, Irmukhamedov A, Andersen M, Borlaug BA, Moller JE. Hemodynamic Characteristics in Significant Symptomatic and Asymptomatic Primary Mitral Valve Regurgitation at Rest and During Exercise. Circ Cardiovasc Imaging. 2018 Feb;11(2):e007171. doi: 10.1161/CIRCIMAGING.117.007171. PMID 29449412
- See also: Related Info — https://open.rsyd.dk/OpenProjects/da/openProject.jsp?openNo=226